CLINICAL TRIAL: NCT04767724
Title: A Prospective Randomized Controlled Clinical Trial Comparing the Extracorporeal Shock Wave and Local Corticosteroid Injection for Carpal Tunnel Syndrome
Brief Title: Extracorporeal Shock Wave Versus Local Corticosteroid Injection for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LH2017-012
Record Dates: First submitted 2021-02-10; First posted 2021-02-23 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Carpal Tunnel Syndrome; Shock Wave
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave (Experimental): Participants received three ESWT sessions once per week for three consecutive weeks. The probe of the ESWT machine (FT-174; Swiss Dolor Class; Switzerland) was placed perpendicularly on the patient's palm over the median nerve on the carpal tunnel after application of the ultrasound gel as a coupling agent. Afterward, the ESWT was administered with 1000 shots, 1.5 bar of pressure, and a frequency of 6 Hz
  Interventions: Device: Extracorporeal shock wave
- Local corticosteroid injection (Active Comparator): A single injection of one mL (40 mg) of betamethasone into the region surrounding the median nerve.
  Interventions: Device: Extracorporeal shock wave

INTERVENTIONS:
Device: Extracorporeal shock wave — Participants received 3 ESWT sessions once per week for 3 consecutive weeks or a single injection of one mL (40 mg) of betamethasone into the region surrounding the median nerve.
  Other Names: Local corticosteroid injection

SUMMARY:
This RCT is to investigate the clinical effect of extracorporeal shock wave therapy (ESWT) compared to the local corticosteroid injection (LCI) in managing mild to moderate carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
To investigate the effect of extracorporeal shock wave therapy (ESWT) compared to the local corticosteroid injection (LCI) in managing mild to moderate carpal tunnel syndrome (CTS). About 50-60 patients with mild to moderate CTS are supposed to be randomly allocated into either ESWT group or LCI group. The outcomes include the visual analog scale (VAS), the Boston Carpal Tunnel Questionnaire (BCTQ), and nerve conduction study at baseline and at 3 weeks, 9 weeks, 12 weeks, 6 months, and 12 months after the treatments.

ELIGIBILITY:
Inclusion Criteria:

The patients aged ≥18 years

1. Should present a new episode of CTS with symptoms lasting for ≥ six weeks
2. Symptoms include wrist pain, numbness, and paraesthesia on the hands
3. Tested postive by the Phalen test and Tinel test
4. Electrodiagnostically diagnosed with mild to moderate CTS

Exclusion Criteria:

1. A lack of consent information
2. A history of a CTS surgery or LCI in the carpal tunnel
3. Asystemic disease that may interfere with the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | At baseline (before the treatment)
  The Visual Analog Scale (VAS) is frequently used as a tool to measure the degree of the pain felt by the participants. The score ranges from 0 to 10. The higher score means a higher degree of the pain.
Visual Analog Scale (VAS) | At 6 months after the treatments
  The Visual Analog Scale (VAS) is frequently used as a tool to measure the degree of the pain felt by the participants. The score ranges from 0 to 10. The higher score means a higher degree of the pain.
Visual Analog Scale (VAS) | At 12 months after the treatments
  The Visual Analog Scale (VAS) is frequently used as a tool to measure the degree of the pain felt by the participants. The score ranges from 0 to 10. The higher score means a higher degree of the pain.
Boston Carpal Tunnel Questionnaire (BCTQ) | At baseline (before the treatment)
  Boston Carpal Tunnel Questionnaire (BCTQ) is the most widely used self-administered outcome scale in patients with carpal tunnel syndrome (CTS) for assessing patients' perceived symptom severity and functional status. The score ranges from 19 to 95. The higher score means a worse status of CTS.
Boston Carpal Tunnel Questionnaire (BCTQ) | At 6 months after the treatments
  Boston Carpal Tunnel Questionnaire (BCTQ) is the most widely used self-administered outcome scale in patients with carpal tunnel syndrome (CTS) for assessing patients' perceived symptom severity and functional status. The score ranges from 19 to 95. The higher score means a worse status of CTS.
Boston Carpal Tunnel Questionnaire (BCTQ) | At 12 months after the treatments
  Boston Carpal Tunnel Questionnaire (BCTQ) is the most widely used self-administered outcome scale in patients with carpal tunnel syndrome (CTS) for assessing patients' perceived symptom severity and functional status. The score ranges from 19 to 95. The higher score means a worse status of CTS.
The peak latency of the median sensory nerve action potential (SNAP) | At baseline (before the treatment)
  The peak latency of the median sensory nerve action potential (SNAP) is used to assess the function status of the median sensory nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The peak latency of the median sensory nerve action potential (SNAP) | At 6 months after the treatments
  The peak latency of the median sensory nerve action potential (SNAP) is used to assess the function status of the median sensory nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The peak latency of the median sensory nerve action potential (SNAP) | At 12 months after the treatments
  The peak latency of the median sensory nerve action potential (SNAP) is used to assess the function status of the median sensory nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The amplitude of the median sensory nerve action potential | At baseline (before the treatment)
  The amplitude of the median sensory nerve action potential is used to assess the function status of the median sensory nerve. The value ranges from 0 μV. The higher value means the better function status of the nerve.
The amplitude of the median sensory nerve action potential | At 6 months after the treatments
  The amplitude of the median sensory nerve action potential is used to assess the function status of the median sensory nerve. The value ranges from 0 μV. The higher value means the better function status of the nerve.
The amplitude of the median sensory nerve action potential | At 12 months after the treatments
  The amplitude of the median sensory nerve action potential is used to assess the function status of the median sensory nerve. The value ranges from 0 μV. The higher value means the better function status of the nerve.
The distal latency of the median compound motor action potential (CMAP) | At baseline (before the treatment)
  The distal latency of the median compound motor action potential (CMAP) is used to assess the function status of the median compound motor nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The distal latency of the median compound motor action potential (CMAP) | At 6 months after the treatments
  The distal latency of the median compound motor action potential (CMAP) is used to assess the function status of the median compound motor nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The distal latency of the median compound motor action potential (CMAP) | At 12 months after the treatments
  The distal latency of the median compound motor action potential (CMAP) is used to assess the function status of the median compound motor nerve. The value ranges from 0 ms. The less value means the quicker conduction of the action potential and the better function status of the nerve.
The amplitude of the median compound motor action potential | At baseline (before the treatment)
  The amplitude of the median compound motor action potential is used to assess the function status of the median compound motor nerve. The value ranges from 0 mV. The higher value means the better function status of the nerve.
The amplitude of the median compound motor action potential | At 6 months after the treatments
  The amplitude of the median compound motor action potential is used to assess the function status of the median compound motor nerve. The value ranges from 0 mV. The higher value means the better function status of the nerve.
The amplitude of the median compound motor action potential | At 12 months after the treatments
  The amplitude of the median compound motor action potential is used to assess the function status of the median compound motor nerve. The value ranges from 0 mV. The higher value means the better function status of the nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Study Chair — Ningbo Medical Center Lihuili Hospital
Locations (1):
- Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang ZJ, China

IPD SHARING:
Plan to Share IPD: Yes
Details of interventions, data of the results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starts on Aug 30, 2019, and will last for 3 years.